CLINICAL TRIAL: NCT06732999
Title: Using Smartphone Sensors to Assess Symptom Relief in Patients With Social Anxiety Disorder Undergoing Gaze Contingent Music Reward Therapy (GC-MRT)
Brief Title: Smartphone Sensors to Assess Symptom Relief in Patients With Social Anxiety Disorder Undergoing Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: BHQ_SA
Record Dates: First submitted 2024-11-24; First posted 2024-12-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-12

CONDITIONS: Social Anxiety Disorder (SAD); Attention; Smartphones; Smartphone Application
Keywords: GC-MRT; Social Anxiety Disorder (SAD); Digital Behaviour; Smartphone; Smartphone assesment
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to three groups with varying intervals between the pre-assessment and the start of treatment, following a multiple-baseline design (Group A - 1 week; Group B - 2 weeks; Group C - 3 weeks). All participants will receive the same treatment (GC-MRT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Starting GC-MRT training after randomized allocation of period of time after assesment (Experimental): Gaze-Contingent Music Reward Therapy (GC-MRT) is a treatment method for adults with social anxiety disorder found to be effective in reducing social anxiety in various RCTs. This method includes a computerized cognitive training to redirect threat-related attention patterns. Time period between Pre assessment and start of GC-MRT is randomly assigned (1 week/ 2 weeks/ 3 weeks) to create a multiple baseline design.
  Interventions: Behavioral: Gaze-Contingent Music Reward Therapy (GC-MRT

INTERVENTIONS:
Behavioral: Gaze-Contingent Music Reward Therapy (GC-MRT — Gaze-Contingent Music Reward Therapy (GC-MRT) is a treatment method for adults with social anxiety disorder found to be effective in reducing social anxiety in various RCTs. This method includes a computerized cognitive training to redirect threat-related attention patterns.

SUMMARY:
The goal of this study is to examine if a digital behavior-based framework, utilizing the BHQ app, can effectively monitor social anxiety symptoms and evaluate the symptom-reducing impact of attentional training for adults (18-65) with social anxiety disorder (SAD), compared to traditional clinical questionnaires and self-reports.

The main questions it aims to answer are:

1. Can the BHQ app provide a reliable digital measure of social anxiety symptoms?
2. Does GC-MRT significantly reduce symptoms of social anxiety as measured through BHQ app monitoring and standard assessment tools?

Researchers will compare the digital BHQ measurements to traditional clinical assessments to see if the app-based measurements is effective in monitoring symptoms relief.

Participants will:

* Complete an initial clinical interview and self-report questionnaires.
* Engage in a computer-based "free-viewing" task for baseline attention assessment using eye tracking.
* Connect to the BHQ app for continuous monitoring throughout the study.
* Undergo attentional training, GC-MRT.
* Complete weekly SPIN assessments.
* Undergo Final evaluation two weeks post-treatment including repeated clinical interviews, self-reports, and the computer-based task to assess changes in attention patterns and symptom reduction.

DETAILED DESCRIPTION:
Research Design The study is a multiple baseline open trial with one active treatment arm and comprises three stages. The interval between the first and second stages varies across groups (one, two, or three weeks) to create a mixed baseline structure. Continuous monitoring via the smartphone App takes place from the first meeting until the final assessment in the third stage.

Stage 1 - Baseline Assessment:

Participants are recruited through social media advertisements (e.g., Google, Facebook) offering participation in a study on a treatment shown to be effective for social anxiety disorder. Potential participants who express interest are invited to an initial clinical assessment following a brief phone screening. Before the assessment, participants are informed of the study process and are asked to provide a written informed consent. A structured clinical interview is then conducted by a trained clinician to evaluate symptom severity and diagnosis and determine eligibility based on the inclusion and exclusion criteria of the study. The evaluation session lasts about two hours and includes:

1. Clinical Interview:

   1.1. MINI (Mini International Neuropsychiatric Interview): A short clinical interview to diagnose major psychiatric disorders in Axis 1 as per DSM-IV and ICD-10 criteria.

   1.2. Clinical Global Impressions (CGI) Scale: Completed by the clinician to assess symptom severity at each evaluation point and to measure improvement relative to baseline at the end of treatment and follow-up.

   1.3. Liebowitz Social Anxiety Scale (LSAS): Structured interview version assessing social anxiety symptoms.
2. Self-Report Questionnaires:

   2.1. Demographic Questionnaire: Includes general background questions on gender, age, country of birth, years of education, academic credentials, ADHD, reading difficulties, current occupation, and treatment history (psychological and pharmacological).

   2.2. Social Phobia Inventory (SPIN): Measures social anxiety symptoms in adults.

   2.3. PHQ-9: Patient Health Questionnaire measuring depression symptoms and functional impairment in adults.

   2.4. GAD-7: Assesses symptoms of generalized anxiety. 2.5. VSAS: this questionnaire is based on the LSAS and assesses social anxiety with images of social scenarios.
3. Free-Viewing Task: This task evaluates eye-gaze patterns toward negative and neutral faces. Participants are shown a 4x4 matrix of faces (16 faces in total) with neutral and disgusted expressions. In each step, participants view a matrix of faces for six seconds. Eye movements are recorded with an eye-tracking device, allowing direct measurement of attention focus on the screen stimuli.
4. The digital monitoring App: Participants are set up to use the App for digital monitoring, which serves as a baseline before treatment begins and is used to assess its impact. Monitoring continues throughout the treatment phase and follow-up assessments.

Stage 2 - Treatment, Symptom Assessment, and App monitoring:

1. Treatment (GC-MRT): The treatment protocol, based on a lab-developed program shown to reduce social anxiety symptoms, includes eight bi-weekly individual sessions over four weeks. Each 30-minute session involves a computerized task that tracks eye movements via eye-tracking, focusing participants' attention away from negative stimuli. During each session, participants choose a music track to play during training, which is played only when they focus on the neutral faces in the matrix. The eye-tracking device records eye movements throughout.
2. Continuous digital behavior monitoring: See description in Section 4.
3. Weekly Self-Report: Participants complete the SPIN (Section 2.2) at the start of each week.

Stage 3 - Post-Treatment Evaluation and Follow-Up:

Approximately two weeks after treatment concludes, participants complete another clinical interview, self-report questionnaires (as described in Stages 1 and 2), and repeat the computerized attention eye-tracking. This stage evaluates the impact of treatment on participants' threat-related attention patterns, as well as symptoms of anxiety and mood. Participants are also informed they may now uninstall the App if they so choose.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected vision, without color blindness.
* A primary diagnosis of social anxiety disorder (based on clinician assessment (LSAS), a MINI interview, and an LSAS score above 50).
* Age range of 18-65.
* Ownership of a smartphone that supports the digital monitoring App.

Exclusion Criteria:

* Prior experience with GC-MRT.
* A current diagnosis of post-traumatic stress disorder (PTSD).
* A current or past diagnosis of psychosis or bipolar disorder.
* Neurological disorder (e.g., epilepsy, brain injury).
* Severe suicidal ideation.
* Substance or alcohol addiction.
* Concurrent treatment (pharmacological or psychosocial).
* Pregnancy.
* Insufficient Hebrew proficiency (unable to complete a clinical interview and/or self-report symptoms and/or perform cognitive tasks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
The Liebowitz Social Anxiety Scale (LSAS) | From Pre meeting measurements in week 0 to post training measurements in week 10
  Clinician-rated severity of social anxiety symptoms

SECONDARY OUTCOMES:
Threat-related attention bias | From Pre meeting measurements in week 0 to post training measurements in week 10
  The proposition of attention allocation to angry vs. neutral faces as measured by a free-viewing task with eye-tracking.
The Social Phobia Inventory (SPIN) | From Pre meeting measurements in week 0 to post training measurements in week 10
  Self-reported severity of social anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, Professor, Principal Investigator — School of Psychological Sciences and Sagol School of Neuroscience, Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arad G, Azriel O, Pine DS, Lazarov A, Sol O, Weiser M, Garber E, Bloch M, Bar-Haim Y. Attention Bias Modification Treatment Versus a Selective Serotonin Reuptake Inhibitor Or Waiting List Control for Social Anxiety Disorder: A Randomized Clinical Trial. Am J Psychiatry. 2023 May 1;180(5):357-366. doi: 10.1176/appi.ajp.20220533. Epub 2023 Mar 22. PMID 36945823